CLINICAL TRIAL: NCT06028347
Title: Phase 1, Randomized, Placebo-Controlled, Observer Blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of an Investigational Self-Amplifying MRNA Influenza Vaccine in Healthy Adults
Brief Title: Safety, Reactogenicity, and Immunogenicity Study of a Self-Amplifying MRNA Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V202_01
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Influenza, Human
Keywords: Influenza; Vaccine; mRNA
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- sa-mRNA vaccine dose 1 (Experimental)
  Interventions: Biological: sa-mRNA vaccine Dose 1
- sa-mRNA vaccine dose 2 (Experimental)
  Interventions: Biological: sa-mRNA vaccine Dose 2
- sa-mRNA vaccine dose 3 (Experimental)
  Interventions: Biological: sa-mRNA vaccine Dose 3
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: sa-mRNA vaccine Dose 1 — self-amplifying mRNA vaccine
  Arms: sa-mRNA vaccine dose 1
Biological: sa-mRNA vaccine Dose 2 — self-amplifying mRNA vaccine
  Arms: sa-mRNA vaccine dose 2
Biological: sa-mRNA vaccine Dose 3 — self-amplifying mRNA vaccine
  Arms: sa-mRNA vaccine dose 3
Biological: Placebo — Saline for injection
  Arms: Placebo

SUMMARY:
This is a Phase 1, first-in-human, randomized, placebo-controlled, observer blind study. The effect of two doses of an investigational vaccine on safety, reactogenicity, kinetics and magnitude of the post-vaccination antibody response will be evaluated at different timepoints as compared to placebo in healthy adults.

Approximately 96 evaluable subjects will be enrolled in this study; n=72 receiving investigational vaccine and n=24 receiving placebo.

The study has a screening period (Day -28 to Day -1), a treatment period (Day 1 to Day 43) and a follow-up period (Day 44 to Day 202).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 18 to 49 years of age OR 65 to 85 years of age, inclusive on the day of informed consent.
2. Individuals with body mass index (BMI) between 18 and 32 kg/m2, inclusive, at screening .
3. Individuals who can comply with study procedures including follow-up .

Exclusion Criteria:

1. Female participants of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of highly effective contraceptive methods from at least 30 days prior to informed consent and who do not plan to do so for the duration of the study.
2. Male participants who have not adhered to using barrier contraception such as a condom during at least 60 days after each vaccination, to prevent semen transfer to their sexual partners and prevent pregnancy of a female partner.
3. Progressive, unstable, or uncontrolled clinical conditions
4. Known hypersensitivity or allergy to any study vaccine component
5. Known history of Guillain-Barré syndrome or other demyelinating disease
6. Condition representing a contraindication to vaccination or blood draw
7. Abnormal function of immune system due to clinical condition, medications, or radiotherapy.
8. Receipt or planning to receive blood products, non-study vaccine, influenza vaccine, mRNA-platform vaccine within different timeframes; previous or from study vaccination.
9. Baseline abnormal clinically significant ECG, laboratory safety parameters or vital signs.
10. Plan to donate blood products (other than for this study), sperm, ova, tissues, or organs up to 60 days following the last vaccination.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with clinically significant abnormal vital signs and/or acute reactions | up to 60 minutes or within 6 hours post vaccination
Number and percentage of subjects reporting reactogenicity: Solicited local and systemic AEs | Day 1 to Day 14 of each post vaccination period
Number and percentage of subjects reporting unsolicited AEs | Day 1 to Day 43
Number and percentage of subjects reporting AEs leading to study withdrawal, Adverse Events of Special Interest (AESIs), medically attended AEs (MAAEs), and serious adverse events (SAEs). | Day 1 to Day 202
Number and percentage of subjects with Grade 3 or greater abnormal clinically significant hematology and chemistry laboratory values | Day 3 to Day 43
Number and percentage of subjects with grading shifts in hematology and chemistry laboratory assessments | Day 3 to Day 43
Serum antibody titer against the HA glycoprotein in terms of GMT, GMFI, and GMT ratio measured via HI assay | Day 1, Day 22, Day 43
Number and percentage of subjects with HAI titer ≥1:10 and <1:10 (lower limit of quantification [LLOQ]) | Day 1, Day 22, Day 43
Number and percentage of subjects with HAI titer ≥1:40, ≥1:80, ≥1:160 and ≥1:320 | Day 1, Day 22, Day 43
Seroconversion rate (SCR) by HAI assay | Day 1, Day 22, Day 43
  SCR defined as the percentage of subjects with either a prevaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40, or a prevaccination HAI titer ≥1:10 and a ≥4-fold increase in post-vaccination

SECONDARY OUTCOMES:
Serum antibody titer against the HA glycoprotein in terms of GMT, GMFI, and GMT ratio measured via HI assay | Day 1, Day 202
Number and percentage of subjects with ≥4-fold increase in post-vaccination HAI titer | Day 1, Day 202
Number and percentage of subjects with HAI titer ≥1:10 and <1:10 (LLOQ) | Day 202
Number and percentage of subjects with HAI titer ≥1:40, ≥1:80, ≥1:160 and ≥1:320 | Day 202
Seroconversion rate (SCR) by HAI assay | Day 1, Day 202
Serum antibody titer against the NA glycoprotein in terms of GMT, GMFI, and GMT ratio measured via ELLA assay | Day 1, Day 22, Day 43, Day 202
Number and percentage of subjects with ≥4-fold increase in post-vaccination ELLA titer | Day 1, Day 22, Day 43, Day 202

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (2):
- Australia (2):
  - Nucleus Network Brisbane Clinic, Brisbane, Queensland
  - Nucleus network Melbourne Clinic, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the CTD modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., ICH E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])).
Supporting Information: Study Protocol, SAP
Time Frame: SEQIRUS discloses results from clinical studies within 12 months of last patient last visit (LPLV) unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication.
URL: http://www.seqirus.us/partnering